CLINICAL TRIAL: NCT02581371
Title: Randomized, Double-blind, Placebo-controlled Study of the Effect of Cerebrolysin® (EVER Neuro Pharma GmbH, Austria) at the Level of Paresis of the Upper Limb When Used in Complex Therapy of Acute Ischemic Stroke
Brief Title: Comprehensive Reparative Therapy in Ischemic Stroke COMplex Repair in Ischemic Stroke-Arm
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Institute of the Brain, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COMRIS-ARM-C
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Ischemic Stroke
Keywords: Cerebrolysin; neuroplasticity; upper limb; middle cerebral artery; NBS; navigation brain stimulation; paretic limb; stroke; ischemic stroke; rehabilitation; Frenchay Arm Test; NBS eXimia Nexstim; Barthel index
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — cerebrolysin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cerebrolysin infusion (Experimental): Cerebrolysin, solution for injection, 10 ml vials. Two 10-day courses of 50 ml of investigational drug + 50 ml of sodium chloride 0.9% iv slowly drip infusions daily, separated with a 7-day interval
  Interventions: Drug: Cerebrolysin infusion
- Placebo infusion (Placebo Comparator): Sodium chloride 0.9%, solution for infusion, 100 ml. Two 10-day courses of 100 ml of sodium chloride 0.9% iv slowly drip daily, separated with a 7-day interval.
  Interventions: Other: Placebo infusion

INTERVENTIONS:
Drug: Cerebrolysin infusion — Two 10-day courses of 50 ml of investigational drug + 50 ml of sodium chloride 0.9% iv slowly drip infusions daily, separated with a 7-day interval
  Other Names: Cerebrolysin
  Arms: Cerebrolysin infusion
Other: Placebo infusion — Two 10-day courses of 100 ml of sodium chloride 0.9% iv slowly drip daily, separated with a 7-day interval
  Other Names: sodium chloride
  Arms: Placebo infusion

SUMMARY:
The aim of the present clinical phase IV study is to estimate the influence of Cerebrolysin in combination with standard therapy on the dynamics of recovery of the paretic upper limb in patients with acute ischemic stroke.

Each patient participates in the study for 176-190 days (approximately 6 months). The estimated duration of the study is 2 years.

DETAILED DESCRIPTION:
Rehabilitation programs and drug therapy in a stroke aimed, primarily, to the stimulation of the processes of neuroplasticity.

After the screening procedures the eligible patients get randomized in 1 of the 2 groups: either the group of a standard therapy in combination with Cerebrolysin infusions, or the group of a standard therapy in combination with placebo infusions.

The therapy consists of the 3 consecutive periods:

1. st - 10 days of daily infusions of Cerebrolysin / placebo;
2. nd - 7 days break;
3. d - 10 days of daily infusions of Cerebrolysin / placebo.

All participants will attend 7 Visits of the study (Visits 0, 1-6) at 2 sites respectively:

1. st - clinical center #1 - Sverdlovsk Regional Clinical Hospital #1, Ekaterinburg
2. nd - clinical center #2 - Clinical Institute of Brain, Ekaterinburg.

Patients will be transferred from the 1st site to the 2nd one at the moment of time between Visit 2 and Visit 3.

Patients will undergo traditional laboratory and clinical examination procedures and several specific ones such as scale NIHSS, modified Rankin scale, Barthel index, hand Frenchy assessments. All hand Frenchy assessments will be videotaped for later evaluation by an authorized researcher.

All participants will undergo the procedure of navigational transcranial magnetic stimulation of the brain NBS eXimia Nexstim with the use of an individual 3D brain model created on the Visit 0 MRI results basis.

Neither the patient nor the doctor will know whether they receive an investigational drug or placebo.

ELIGIBILITY:
Inclusion criteria:

1. A signed patient informed consent;
2. Men and women at the age from 45 years to 75 years, inclusive;
3. Confirmed (clinically and by MRI of the brain) diagnosis of acute ischemic stroke in the basin of the middle cerebral artery;
4. The severity of the stroke from 5 to 24 points on a scale NIHSS;
5. Hemiparesis, mainly affecting the upper limbs (not more than 2 points in the evaluation function of the affected hand using the test for hand Frenchay and not more than 2 points in the evaluation of the affected lower limb 6-point scale NIHSS);
6. The time from the onset of the disease prior to the introduction of the drug for 72 hours;
7. The willingness of patients of both sexes and their sexual partners with preserved reproductive function to use reliable methods of contraception, starting from the moment of inclusion in the study until the completion of participation in this clinical study.

Exclusion Criteria:

1. The age of 45 years or older than 75 years;
2. Known intolerance (including allergic reactions) Cerebrolysin, excipients of the investigational medication;
3. Thrombolytic therapy;
4. Signs of a hemorrhagic stroke;
5. Impairment of consciousness (≥ 2 points during the evaluation under item 1A NIHSS);
6. The presence of elements allowing to predict the resolution of neurological symptoms within 24 hours from the first symptoms;
7. Stroke or transient ischemic attack in history;
8. The score on the modified Rankin scale to a stroke more than 0 points;
9. Concomitant therapy or neuroprotective nootropic drugs;
10. New-onset seizures or epilepsy;
11. Planned carotid endarterectomy or other operations for secondary prevention of stroke;
12. Neurological disease or pathology of the neuromuscular system or any other disease that may affect the interpretation of study results;
13. Systemic therapy with biological drugs, including interferon, inductors and/or cytokine/anti-cytokine (e.g., anti-TNF, anti-CD4, IL-10, IL-1, etc.) within 1 month prior to screening;
14. Severe concomitant diseases, including cancer, which, in the opinion of the investigator, may affect the estimated parameters;
15. Uncontrolled hypertension (SBP ≥ 220 mm Hg. CL. and/or DBP ≥ 120 mm Hg. article in repeated measurements at the screening visit);
16. Uncontrolled angina, congestive heart failure or severe arrhythmia;
17. The presence of chronic infection (hepatitis B, C or AIDS) in the active form.
18. Severely impaired renal function or hepatic impairment (total bilirubin no more than 1.5 hvgn, the level of serum creatinine no more than 2.5 hugn and the levels of ALT, AST, GGT is not higher than 2.5 hvgn);
19. Diseases of the blood;
20. Mental illness, severe depression or suicide attempts in history;
21. The a history of drug addiction, alcoholism and abuse of drugs;
22. Contraindications to MRI: metal body, splinters, ferromagnetic implants (pacemakers, automatic dosing of drugs, implanted insulin pumps, artificial anus with a magnetic closure, artificial heart valves with metal elements), steel implants (clamps/clips on blood vessels, artificial joints, metal osteosynthesis devices), hearing AIDS;
23. Participation in any other clinical study within 30 days prior to screening or simultaneous participation in other clinical studies;
24. Pregnancy, breastfeeding or planning a pregnancy;
25. Women and men with preserved reproductive potential who refuse to use effective methods of contraception throughout the study;
26. Life expectancy less than 1 year;
27. Any disease or circumstances that, in the opinion of the investigator, may interfere with the subject participating in the study or in relation to which participation in the study may be dangerous for the subject;

Premature withdrowal criteria:

1. The research subject may discontinue participation at any time without giving a reason;
2. The researcher ahead of time to exclude the patient from the study in the following cases;
3. The refusal of the subject from further participation in the study;
4. Failure to comply with the subject rules of participation in the study;
5. The reasons that emerged during the study and threatening the security of the subject, including those associated with taking study medication adverse events;
6. The entities with during the study pregnancy;
7. The application of the patient in the study period of any additional neuroprotective and nootropic drugs, drugs from the group of correctors of cerebral blood flow;
8. Other reasons arising in the course of the study and prevent the realization of the study according to the Protocol;
9. Repeated stroke in the course of the study;
10. Subjects who are lost to observation, also belong to prematurely withdrawn from the study.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Overall dynamics of the hand function assessed by the Frenchay Arm Test | 6 months
  Visit 5 data comparison with Visit 0 data

SECONDARY OUTCOMES:
Dynamics of the hand function assessed by the Frenchay Arm Test | 6 months
  Visits 2,3,4 data comparison with Visit 0 data
Dynamics of the grades on the NIHSS scale | 6 months
  Visits 2,3,4,5 data comparison with Visit 0 data
Dynamics of the grades on the modified Rankin scale | 6 months
  Visits 2,3,4,5 data comparison with Visit 0 data
Dynamics of the Barthel index changes | 6 months
  Visits 2,3,4,5 data comparison with Visit 0 data
Dynamics of the cerebral infarction volume decrease according the 3D MRI data | 6 months
Dynamics of the hemispheres cortex topology of palms motor centers according to navigated transcranial stimulation of the brain (NBS) | 6 months
  Visit 4, 5 data comparison with Visit 3 data
Dynamics of motor response threshold based on the results of navigated transcranial stimulation of the brain (NBS) | 6 months
Dynamics of the amplitude of motor responses | 6 months
Dynamics of the latency of motor responses | 6 months
Frequency, nature and severity of adverse events. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Avgustovich Belkin, Prof.,MD,PhD, Study Director — Clinical Institute of Brain
Locations (2):
- Russia (2):
  - Clinical Institute of Brain, Beryozovsky, Sverdlovsk Oblast
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg, Sverdlovsk Oblast

REFERENCES:
- See also: Clinical Institute of Brain. Official website — http://www.neuro-ural.ru/
- See also: Sverdlovsk Regional Clinical Hospital #1. Official website — http://www.okb1.ru